CLINICAL TRIAL: NCT05457803
Title: Real-world Momentary Assessment of Kratom Use Accompanied by Product Assays: A Natural-history Study for Interdisciplinary Characterization of Kratom Use and Pharmacology
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000910; 000910-DA
Record Dates: First submitted 2022-07-13; First posted 2022-07-14 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07-02

CONDITIONS: Chronic Pain; Fatigue; Substance Use Disorders
Keywords: Alkaloid Content; Mitragyna Speciosa; Mitragynine; 7-Hydroxymitragynine; Corynoxine; Speciociliatine; As Serotonergic, Dopaminergic, Adrenergic, And Adenosinergic Receptors; Natural History
MeSH Terms: conditions — Chronic Pain; Fatigue; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- In-persom kratom users: 10 subjects that use kratom an additional cross-sectional evaluation: one session day at the NIDA IRP preceded by a consent session day; 2 visits at our BRC building total.
- Online kratom users: 240 subjects that use kratom, prospective observational cohort study in which each participant provides intensive longitudinal data on kratom use for 15 consecutive days via smartphone app

SUMMARY:
Background:

Mitragyna speciosa, also called kratom, is a plant used in Southeast Asia for its psychoactive effects. Its use has increased in the US, and an estimated 10 million adults may take it at least semiregularly. Most scientific research on human use of kratom has consisted of surveys in which people looked back on their experiences with it. Results from those surveys have been useful, but, like many behaviors, kratom use can be more fully understood if it is also studied as it happens. The technical term for this procedure is ecological momentary assessment (EMA). In EMA, people report their moods and activities in real time, a few times per day, usually with a smartphone app.

Objective:

This natural history study will collect data about how people use kratom and how it affects them.

Eligibility:

People aged 18 and older who use kratom 3 or more times per week

Design:

Most participants will be remote only.

They will fill out an online consent form. They will also answer an initial set of questions about their kratom use.

They will download an app on their smartphones for EMA (described above). They will use this app to answer short sets of questions for 15 days in a row about their ongoing behaviors and moods, including kratom use.

They will use a prepaid envelope to mail in a sample of their kratom product.

Some participants, after doing the EMA part of the study, can also come to a clinic. They will have 1 visit for informed consent (1-3 hours) and 1 visit for a monitoring session (8 hours) where we can directly assess the effects of their usual dose of kratom. They will bring their kratom produce with them to take on site.

Before they take the kratom, they will have a physical exam. They will have blood and urine tests. They will answer questions about their sleep, driving, and general feelings. They will complete tasks on a computer to measure their reflexes and response times. Their driving performance will be assessed in a simulator.

Researchers will watch participants consume their kratom. A sample of their product will be taken for analysis.

After taking their kratom, those participants will repeat some questionnaires and tests, including the driving simulation. They will also be interviewed about their use of kratom....

DETAILED DESCRIPTION:
Study Description:

Our natural-history study will build on preliminary research on the use and effects of kratom. We propose to examine momentary reasons for and self-reported effects of kratom-product use in daily life, associations of these findings with product alkaloid content and, in a direct-observation setting, externally observable effects of kratom-product use.

In the Main EMA Study, to be conducted nationwide via online/mobile data collection, we will examine instances of kratom use in naturalistic settings using EMA, and we will characterize the alkaloid content of the products used. The target sample size is 240 completers.

In the In-person Substudy, 10 participants who reside near the NIDA IRP will conduct the same activities as in the Main EMA Study (online questionnaires, then EMA for 15 days), plus a one-day outpatient session. On the session day, we will collect physiological and task-derived measures (these will include a driving-simulation task) after the participants have taken their regular kratom product dose. This will be followed by semi-structured narrative qualitative interviews.

Objectives for the Main EMA Study:

Primary objective: to collect momentary assessments of individual instances of kratom use and effects associated with use (e.g., sleep duration, mood, motivations for use, acute effects, etc.) in daily life over 15 days among regular kratom users, for better understanding kratom use in real-world contexts and in real time.

Secondary objective: to determine associations of momentary responses with directly assayed content of samples of participants kratom products.

Exploratory objectives: to evaluate whether retrospective self-report on cross-sectional questionnaires completed prior to EMA correlate with momentary self-report (e.g., do people who report using kratom primarily for pain actually report self-treatment of pain symptoms as a proximal motivation?). A second exploratory objective is to determine whether there are subgroups of participants who share distinct patterns of kratom use.

Objectives for the In-Person Substudy:

Primary objective: to evaluate the relationships among subjective self-reported kratom effects (measured over 3 hours post-dosing), the kratom product used, and kratom alkaloid concentrations in biospecimens.

Secondary objective: to gather comprehensive narrative case-report data via qualitative interviewing.

Exploratory objectives include: First, to assess vital signs, pupil size, and psychomotor performance of participants prior to their taking their regular kratom dose and at repeated intervals subsequent to their taking their regular kratom product dose (4-6 total time points). Second, to measure signs of opioid withdrawal among participants prior to their taking their regular kratom dose and after (4 total time points). Third, to measure participants performance on a driving simulation before they have taken their kratom dose and after they have taken their kratom dose (2 time points total).

Endpoints for Main EMA Study:

For primary objectives: proximal motivations for use; somatic and psychoactive effects reported from use; associations between self-reported states (e.g., mood, pain, craving), and particular kratom product types reported as being used; associations between self-reported states (e.g., mood, pain, craving) and kratom dose.

For secondary objectives: quantification of up to 14 kratom alkaloids; differences in alkaloid content by kratom product type (e.g., extract, raw plant matter); differences in alkaloid content by kratom vendor type (e.g., small online vendor, large-scale importer and distributor; between-person correlations (self-reported momentary effects and alkaloid levels).

For exploratory objectives: correlation of cross-sectional self-reported kratom use motivations and momentary (proximate) kratom use motivations; Cluster analysis of kratom use patterns.

Endpoints for In-person Substudy:

For primary objectives: Concentrations of detectable kratom alkaloids and their metabolites in human plasma and urine; differences in concentrations by kratom product type (e.g., extract, raw plant matter); Addiction Research Center Inventory and other self-report questionnaires.

For secondary objective: narrative case report series documenting participant s kratom use, from initiation to present day.

For exploratory objectives: Psychomotor performance; Resting vitals; Pupil size; Subjective Opioid Withdrawal Scale; Driving-simulation performance.

ELIGIBILITY:
* INCLUSION CRITERIA:

For the Main EMA Study

* Regular kratom use.
* Passing data validity checks on the online screening questionnaire.
* Reporting ownership of a smartphone.
* Age >= 18 years.
* Currently residing in the US .
* Willingness to complete all study activities as described in the online study preamble and informed consent, including willingness to provide a small sample of their kratom product.
* Passing online Main Study consent quiz with at least 8/10 correct answers.
* English language proficiency.
* Not incarcerated.

Additional inclusion criterion for the In-person Substudy:

-Residing in or near MD.

EXCLUSION CRITERIA:

For the Main EMA Study

* Missing data validity checks on screening questionnaire
* Decisionally impaired adults..

Additional exclusion criterion for the In-person Substudy:

* Pregnancy by urine test.
* Self-reported proneness to experiencing motion sickness or feelings of vertigo. This is a precaution, because motion sickness could interfere with the task or cause discomfort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Main EMA Study the subjects will be selected online form subjects who use kratom ( Target 240 completers). For the In-person Substudy (target 10 subjects) we will select online or local form subjects who use kratom.
Sampling Method: Non-Probability Sample
Enrollment: 396 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
motivations for use of kratom | End of study
  To collect momentary assessments of individual instances of kratom use and effects associated with use (e.g., sleep duration, mood, motivations for use, acute effects, etc.) in daily life over 15 consecutive days among regular kratom users, for better understanding of kratom use in real-world contexts and in real time.
Differences in concentrations by kratom product type | End of study
  To evaluate the relationships among subjective self-reported kratom effects (measured over 3 hours post-dosing), the kratom product used, and kratom alkaloid concentrations in biospecimens.
Associations between self-reported states and particular kratom product types reported as being used. | End of study
  To collect momentary assessments of individual instances of kratom use and effects associated with use (e.g., sleep duration, mood, motivations for use, acute effects, etc.) in daily life over 15 consecutive days among regular kratom users, for better understanding of kratom use in real-world contexts and in real time.
Somatic and psychoactive effects reported from use of kratom | End of study
  To collect momentary assessments of individual instances of kratom use and effects associated with use (e.g., sleep duration, mood, motivations for use, acute effects, etc.) in daily life over 15 consecutive days among regular kratom users, for better understanding of kratom use in real-world contexts and in real time.
Associations between self-reported states and kratom dose | End of study
  To collect momentary assessments of individual instances of kratom use and effects associated with use (e.g., sleep duration, mood, motivations for use, acute effects, etc.) in daily life over 15 consecutive days among regular kratom users, for better understanding of kratom use in real-world contexts and in real time.
Detect Concentrations of detectable kratom alkaloids and their metabolites in human plasma and urine. | End of study
  To evaluate the relationships among subjective self-reported kratom effects (measured over 3 hours post-dosing), the kratom product used, and kratom alkaloid concentrations in biospecimens.
Complete addiction Research Center Inventory (ARCI). | End of study
  To evaluate the relationships among subjective self-reported kratom effects (measured over 3 hours post-dosing), the kratom product used, and kratom alkaloid concentrations in biospecimens.

SECONDARY OUTCOMES:
Evaluate Psychomotor performance, Resting vitals, Pupil size, Drug Effects Questionnaire, Subjective Opioid Withdrawal Scale (SOWS), Driving-simulation performance. | End of study
  To assess vital signs, pupil size, and psychomotor performance prior to their taking their regular kratom dose and at repeated intervals subsequent to their taking their regular kratom dose (4-6 total time points). To measure signs of opioid withdrawal among participants prior to their taking their regular kratom dose and after (6 total time points). To measure participants performance on a driving simulation before they have taken their kratom dose and after they have taken their kratom dose (2-time points total).
Correlation of cross-sectional self-reported kratom use motivations and momentary (proximate) kratom use motivations. | End of study
  To evaluate whether retrospective self-report on cross-sectional questionnaires completed prior to EMA correlate with momentary self-report (e.g., do people who retrospectively report using kratom primarily for pain actually report self-treatment of pain symptoms as a proximate motivation?). To determine if there are subgroups of kratom user within the larger sample
Quantification of up to 14 kratom alkaloids | End of study
  To determine associations of momentary responses with directly assayed content of samples of participants kratom products.
Use-pattern clusters | End of study
  To evaluate whether retrospective self-report on cross-sectional questionnaires completed prior to EMA correlate with momentary self-report (e.g., do people who retrospectively report using kratom primarily for pain actually report self-treatment of pain symptoms as a proximate motivation?). To determine if there are subgroups of kratom user within the larger sample
Between-person correlations (self-reported momentary effects and alkaloid levels). | End of study
  To determine associations of momentary responses with directly assayed content of samples of participants kratom products
Narrative case report series documenting participants kratom use, from initiation to present day | End of study
  To gather comprehensive narrative case report from participants via qualitative interviewing.
Differences in alkaloid content by kratom vendor type | End of study
  To determine associations of momentary responses with directly assayed content of samples of participants kratom products
Differences in alkaloid content by kratom product type | End of study
  To determine associations of momentary responses with directly assayed content of samples of participants kratom products.

CONTACTS AND LOCATIONS:
Overall Officials: David H Epstein, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

REFERENCES:
- [Background] Berthold EC, Kamble SH, Raju KS, King TI, Popa R, Sharma A, Leon F, Avery BA, McMahon LR, McCurdy CR. Preclinical pharmacokinetic study of speciociliatine, a kratom alkaloid, in rats using an UPLC-MS/MS method. J Pharm Biomed Anal. 2021 Feb 5;194:113778. doi: 10.1016/j.jpba.2020.113778. Epub 2020 Nov 21. PMID 33277117
- [Background] Anwar M, Law R, Schier J. Notes from the Field: Kratom (Mitragyna speciosa) Exposures Reported to Poison Centers - United States, 2010-2015. MMWR Morb Mortal Wkly Rep. 2016 Jul 29;65(29):748-9. doi: 10.15585/mmwr.mm6529a4. PMID 27466822
- [Background] Babu KM, McCurdy CR, Boyer EW. Opioid receptors and legal highs: Salvia divinorum and Kratom. Clin Toxicol (Phila). 2008 Feb;46(2):146-52. doi: 10.1080/15563650701241795. PMID 18259963